CLINICAL TRIAL: NCT06844565
Title: Role of IL 12 and IL 23 as Potential Biomarkers in Diagnosis of Early Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Galal Flefel, Lecturer of Internal Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264PR1059/1/25
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Interleukin 12; Interleukin 23; Biomarker; Diagnosis; Crohn Disease
MeSH Terms: conditions — Disease; Crohn Disease | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients who are suspected of having Crohn's disease clinically and by colonoscopy (like ulcers, fistulas, or skip lesions). Non-specific ileitis by histopathology.
  Interventions: Procedure: Immunohistochemistry procedure

INTERVENTIONS:
Procedure: Immunohistochemistry procedure — Briefly, all slides will be rehydrated, and antigen retrieval will be performed using sodium citrate (pH = 6.0) in a pressure cooker (EDTA buffer, pH = 8.4).
  All slides will be blocked with endogenous peroxidase with 3% hydrogen peroxide and blocked non-specific protein with 2.5% bovine serum albumin in phosphate-buffered saline.
  If the result shows non-specific ileitis, immunohistochemical staining for IL-12 and IL-23 will be performed using sandwich enzyme-linked immunosorbent assays (ELISA).

SUMMARY:
This study aims to evaluate the role of Interleukin (IL)-12 and IL-23 as potential biomarkers in the diagnosis of early Crohn's disease.

DETAILED DESCRIPTION:
Crohn's disease (CD) is characterized by periods of remission and relapse, with symptoms ranging from abdominal pain and diarrhea to severe complications such as fistulas and intestinal obstruction.

Interleukins (ILs) are known clusters of cytokines that regulate the proliferation, development, and activation of immune cells. IL-12 is predominantly a pro-inflammatory cytokine secreted by antigen-presenting cells (APC) in response to sensing of microbial components by Toll-like receptors. Another member of this family, IL-23 is also produced by DCs and macrophages after toll-like receptors (TLRs) engagement.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* Patients who are suspected of having Crohn's disease clinically and by colonoscopy (like ulcers, fistulas, or skip lesions).
* Non-specific ileitis by histopathology.

Exclusion Criteria:

* Patients with no pathological samples through colonoscopy.
* History of other significant gastrointestinal diseases (e.g., colon cancer, ischemic bowel disease).
* Immunosuppressive therapy or biologic agents at the time of study.
* Previous abdominal surgeries.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study will be carried out on 110 patients suspected of having Crohn's disease are present in Tanta University Hospitals in the period from January 2021 to December 2023 and the data will be collected in the duration from February 2025 to May 2025 that after approval from the institutional ethical committee.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity of IL-23 to predict Crohn's disease | 6 months after procedure
  Sensitivity of IL-23 to predict Crohn's disease will be recorded.

SECONDARY OUTCOMES:
Sensitivity of IL-12 to predict Crohn's disease | 6 months after procedure
  Sensitivity of IL-12 to predict Crohn's disease will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.